CLINICAL TRIAL: NCT03241043
Title: Single Center, Open-label, Randomized, Controlled, Cross Over Study to Evaluate the Pharmacokinetic and Bioavailability of Envarsus® in Comparison to Advagraf® in de Novo Liver Transplant Recipients
Brief Title: Study to Evaluate Pharmacokinetic and Bioavailability of Envarsus® vs. Advagraf® in Liver Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PAKT CTC 151043
Record Dates: First submitted 2016-09-12; First posted 2017-08-07 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Liver Transplantation
Keywords: Pharmacokinetic study; Comparing Envarsus versus Advagraf
MeSH Terms: interventions — Therapeutics; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Envarsus - Advagraf (Experimental)
  Interventions: Drug: Treatment 2 weeks Envarsus followed by 2 weeks Advagraf
- Advagraf - Envarsus (Active Comparator)
  Interventions: Drug: Treatment 2 weeks Advagraf followed by 2 weeks Envarsus

INTERVENTIONS:
Drug: Treatment 2 weeks Envarsus followed by 2 weeks Advagraf
  Arms: Envarsus - Advagraf
Drug: Treatment 2 weeks Advagraf followed by 2 weeks Envarsus
  Arms: Advagraf - Envarsus

SUMMARY:
Single centre, open-label, randomized, controlled, cross over study to evaluate the pharmacokinetic and bioavailability of Envarsus® in comparison to Advagraf® in de novo liver transplant recipients

DETAILED DESCRIPTION:
Using an open-label, randomized, controlled, 2-period cross-over design, two treatments (Envarsus® and Advagraf®) will be compared (with regard to PK profile and bioavailability) after administration of IMP to 20 de novo transplanted recipients. The patients will be randomly assigned to one of the two treatments as treatment period 1 and afterwards switched to treatment period 2 (Group 1: Envarsus® - Advagraf®; Group 2: Advagraf® - Envarsus®).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the patient information and to personally sign and date the informed consent to participate in the clinical trial, before completing any clinical trial related procedures.
2. Male or female recipients ≥ 18 years of a liver graft from a deceased or living donor
3. The patient must receive a twice daily Tacrolimus based immunosuppression treatment.
4. Females of child-bearing potential who agree to comply with any applicable contraceptive requirements of the protocol or females who are permanently sterilized (at least 6 weeks post sterilization).
5. Non-pregnant, non-lactating female.
6. Recipients of a first or re-liver transplant in the last 30 days
7. The patient is co-operative and available for the entire clinical trial.

Exclusion Criteria:

1. Patients with a known hypersensitivity to any of the drugs used in the study.
2. Patients who are not able to take oral medication at the time point of randomization.
3. Recipients of combined organ transplants.
4. Patients who are recipients of AB0 incompatible transplant grafts.
5. Currently participation in a clinical trial and any IMP intake within the last four weeks.
6. Patients who use drugs known to strongly interact with the cytochrome P-450 3A4 pathway and therefore influence the tacrolimus blood level are not allowed during Envarsus®/Advagraf® treatment period.
7. Patient with renal impairment with need of dialysis treatment at the time point of randomization.
8. Patient with a quick value < 30 %
9. Patient with a thrombocytopenia <20 Mrd./L
10. Patients with a leukopenia < 1.0 Mrd. / L
11. Patients with inability of oral food intake.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
DAV (average cumulative dose) = cumulative dose per study period/ period days | 20 month
C0/doses (trough level at steady state / daily dose at steady state) | 20 month
AUC0-24/doses | 20 month

CONTACTS AND LOCATIONS:
Overall Officials: Herden, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Hospital Hamburg-Eppendorf, Hamburg, Germany